CLINICAL TRIAL: NCT06367569
Title: Multicenter Evaluation of Baseline MRI Screening With Extended Follow-up of Pineal Cysts for Early Detection of Pineoblastoma in Children With Retinoblastoma
Brief Title: Evaluation of MRI of the Pineal Gland in Retinoblastoma
Acronym: TRbFU
Status: Completed | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Marcus de Jong, Principal investigator, Amsterdam UMC, location VUmc
Other Study IDs: 2012//375
Record Dates: First submitted 2024-04-04; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Retinoblastoma
MeSH Terms: conditions — Retinoblastoma | interventions — Mass Screening; Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Screening for trilateral retinoblastoma with MRI — The diagnostic accuracy of the screening program, baseline screening with MRI followed by follow-up of suspicious pineal glands in heritable retinoblastoma patients.

SUMMARY:
Rationale: Currently baseline brain MRI (magnetic resonance imaging) with extended follow-up of pineal cysts is systematically performed in all new retinoblastoma (Rb) patients, because children with hereditary retinoblastoma have an increased risk of primitive neuroectodermal tumors (PNET) that are histopathologically identical to the retinal tumors (1). The prevalence of developing a PNET in combination with unilateral or bilateral hereditary Rb is 5-15% (2). Treatment is difficult and the prognosis is poor as only few survivors are reported. Only patients with small asymptomatic PNETs (<15 mm) are potentially curable.

Objective: The main objective of this prospective multicenter study is to evaluate the current strategy of baseline MRI screening of the brain in newly diagnosed retinoblastoma patients, with extended follow-up of selected patients with simple and complicated pineal cysts.

Study design: The investigators propose a prospective cohort study (part of a larger multicenter study) to investigate the diagnostic accuracy and survival of baseline MRI screening of the pineal gland in new patients with retinoblastoma, with extended follow-up of selected patients with pineal cysts for early detection of pineoblastoma.

Study population: Within the European Retinoblastoma Imaging Collaboration (ERIC) about 150 new retinoblastoma patients are diagnosed every year. About 10 percent of all new retinoblastoma patients will be diagnosed at the VUmc. According to our sample size calculations the investigators will need 334 Rb patients.

Main study parameters/endpoints: The primary endpoint of the study is pineoblastoma or supra- / parasellar PNET on MRI (index test). Because a gold standard will not be available, tumor cells in cerebrospinal fluid, histopathological confirmation, clinical disease progression during follow-up, and/or follow-up MRI diagnostics will be used as a composite reference standard in case of a positive index test and clinical diagnosis of pineoblastoma or supra- / parasellar PNET within one year of the last MRI will be used as a composite reference standard in case of a negative index test.

DETAILED DESCRIPTION:
1. INTRODUCTION AND RATIONALE Currently baseline brain MRI with extended follow-up of pineal cysts is systematically performed in all new retinoblastoma patients since children with hereditary retinoblastoma have an increased risk of primitive neuroectodermal tumors (PNET) that are histopathologically identical to the retinal tumors. This combination is also known as trilateral retinoblastoma (TRb). The prevalence of developing a PNET in combination with unilateral or bilateral hereditary retinoblastoma is 5-15%. The risk of developing TRb in Rb patients, is less than 0.5% for sporadic unilateral disease. The PNET usually arises in the pineal gland (PG) (77%) but can also be a parasellar or suprasellar tumor. A meta-analysis from 1999 including TRb patients from literature covering 1966 to 1998; they found that the interval between the ocular tumor and the intracranial tumor was 1 versus 22 months respectively in TRbs diagnosed in patients with screening versus patients who developed symptoms. Of TRb cases found at screening half were present when Rb was diagnosed and that 75% might be detected within one year after Rb diagnosis. Treatment is difficult and the prognosis is poor as only few survivors are reported. In a previous retrospective multicenter study from the ERIC-group small asymptomatic PNETs (<15 mm), that were present synchronously with the eye cancer (on baseline MRI) showed to have a better prognosis. Furthermore it was discovered that the majority of early stage pineoblastoma showed a cystic aspect, sometimes hardly distinguishable from benign pineal cysts (9,11,12). The prevalence of pineal cysts in hereditary Rb patients is 5.3%. In the general population at an age of 1 to 5 years 1.6% (1.1% in males and 2.2% in females) of all patients have pineal cysts. Current practice is based on evidence that early depiction of TRbs in retinoblastoma patients (during baseline MRI and follow-up of selected patients with pineal cysts) detects these aggressive tumors in a curable stage.
2. OBJECTIVES The main objective of this prospective multicenter study is to evaluate the current clinical strategy of baseline MRI screening of the brain in newly diagnosed retinoblastoma patients, with extended follow-up of selected patients with simple and complicated pineal cysts.

To investigate this objective the investigators will try to answer the following question: "What is the diagnostic accuracy (sensitivity and specificity) of the baseline MRI screening and extended follow-up of patients with pineal cysts for the diagnosis of TRb?" and: "How can the investigators optimize this screening strategy in order to minimise patient burden by keeping number of MRIs to a minimum and to maximise diagnostic accuracy?" The investigators will evaluate the classification (see section 3.7) of pineal cysts (probably benign versus suspicious) and pineoblastoma or supra- / parasellar PNET.

2.1 Secondary objectives

1. Evaluate epidemiological parameters:

   1. incidence of TRb patients at baseline MRI (synchronous), follow-up (metachronous) MRI, and missed by MRI, compared to historical data;
   2. survival of patients with positive TRb findings on MRI at baseline or follow-up compared to TRb patients missed by MRI and compared to historical data.
2. Evaluate prognostic parameters (age, tumor size, aspect, time of diagnosis relative to Rb diagnosis etc).
3. STUDY DESIGN The investigators propose a prospective multicenter cohort study (to investigate the diagnostic accuracy of baseline MRI screening of the pineal gland in new patients with retinoblastoma, with extended follow-up of selected patients with pineal cysts for early detection of pineoblastoma.

3.1 Study population Within ERIC about 150 new retinoblastoma patients are diagnosed every year. About 10 percent of all new retinoblastoma patients will be diagnosed at the VUmc.

3.2 Inclusion criteria

* All new hereditary and non-hereditary retinoblastoma patients undergoing a baseline MRI diagnosed at one of the ERIC centers.
* Availability of MR sequences (see section 3.7.1) required by the study

3.3 Exclusion criteria

A patient will be excluded from the study if:

* baseline MRI has not been performed;
* MR protocol or quality not adjusted to the required protocol
* Follow-up not possible or available

3.4 Study quality In 2003 The STARD (standards for the reporting of diagnostic accuracy studies) statement has been published by Bussuyt et al. as a tool to help researchers to improve the accuracy and completeness of reporting of studies of diagnostic accuracy. This should allow readers to assess internal validity (potential bias) and external validity (generalisability) of a study. The investigators will use STARD to ensure that - where possible - the design of this study meets those standards and that the final publication is clear on possible risk of bias and generalisability.

3.5 Sample size calculation In the VUmc and the other ERIC centers 150 new retinoblastoma patients are diagnosed each year. All new Rb patients receive a baseline MRI for (clinical) diagnostic purposes. When a pineal cyst is detected on baseline MRI a follow-up MRI will be done (see section 3.7 for the follow-up protocol). The investigators consider the baseline MRI and the follow-up MRI as one diagnostic test (the index test) and the investigators will calculate sample sizes based on that. As mentioned in section 1. 75% of TRb cases can be diagnosed during follow-up within one year, of which 50% can be diagnosed synchronously with Rb. The other 25% of cases develop at a later stage; the investigators will not consider those as false negatives of our test. There are no previous studies on diagnostic accuracy on comparable tests, but on the basis of clinical experience the investigators estimate a sensitivity of at least 95% and a specificity of about 80%. Prevalence in the hereditary Rb group (40% of patients) is about 10, giving us a prevalence of four per cent.

Sensitivity depends on the number of cases; therefore the investigators calculate the needed number of cases according to the estimated sensitivity of 95%. The sample size the investigators calculate has a probability of at least 85% (1 - β) that the 95% (1 - α) lower confidence limit is ≥ 60%. These input variables result in a required number of cases of ten. Entering the number of cases in the previously mentioned formula gives us 240 controls. The investigators can then calculate the 95% lower confidence limit of the expected specificity of 80%. With a probability of at least 85% this number of controls gives us a 95% lower confidence limit of ≥ 72.

The number of required Rb patients is 240 controls + 10 cases = 250, and since 75% of TRb cases can be diagnosed in the first year the investigators need 334 Rb patients for this study. About 10% of Rb patients included in this study will be from the VUmc. The investigators expect almost all Rb patients to participate in the study. With a study duration of about two to three years the investigators expect to be able to include the required number of Rb patients. This sample size calculation is based on rough estimates and could therefore vary. Because of the low number of cases it is especially important to obtain a sufficient number of TRb cases for this study and depending on the number of found cases the duration of this study may vary.

The prevalence of pineal cysts in hereditary Rb patients is about 5% and the investigators estimate the prevalence of pineal cysts in the non-hereditary group is similar to the general population, which is about 1.6%. These numbers amount to (5.3% • 40% + 1.6% • 60%) • 334 = 10 patients with a pineal cyst who will receive follow-up MRIs.

3.6 Study procedures

The ERIC guideline for imaging retinoblastoma states that brain screening for pineoblastoma should be performed in every new patient with retinoblastoma (uni- and bilateral). Pineal lesions depicted on baseline MRI are classified as:

1. normal pineal gland; no further follow-up;
2. probably benign pineal cyst; this group contains patients with a cystic pineal gland with a discrete rim enhancement and a thin smooth wall. Pineal glands with thin intracystic septa will also be classified as probably benign pineal cysts. Follow-up MR imaging will be done once after 3 months and further follow-up is not necessary if the cysts remains stable*;
3. suspicious pineal cyst; irregularly thickened (> 2 mm) cyst wall or fine nodular aspect of the wall. MRI follow-up also after 3 months. If stable, no further follow-up. If any doubt persists, another follow-up after 3 months*;
4. pineoblastoma or supra- / parasellar PNET.

   * In case a patient receives chemotherapy a scan 3 months after chemotherapy is done, to exclude a possible chemotherapy effect on the PNET growth.

3.6.1 MRI protocol This screening is primarily achieved by a post-contrast 3D T1-weighted sequence with 1 mm slice thickness or post Gadolinium thin slice (≤3mm) T1-weighted. The preferred sequence for initial evaluation and follow-up are thin slice (≤ 3mm) T2-weighted (T2-TSE or CISS-images). Follow-up should be performed with the same T2-weighted and post-contrast 3D-T1 weighted sequence.

3.7 Follow-up of subjects withdrawn from treatment Survival data and disease progression will be followed up in all included Rb patients.

4. STATISTICAL ANALYSIS Sensitivity and specificity will be the main measures of outcome of this study. The low number of expected TRb cases will probably not allow for subset analyses. The diagnostic index test the investigators are evaluating (the baseline MRI and the follow-up MRI) lacks a uniform reference standard, however, it is possible to construct a composite reference standard. For positive index test results it might be difficult to determine false positives in some cases, because in case of a positive index test treatment will have been started, which could make it hard to distinguish effect of treatment from a false positive index test result, when a reference test is carried out at a later stage than the MRI. A good reference standard is especially critical for patients where MRI results are not clear cut. See table 1 for the expected test results based on the data the investigators used in our sample size calculation (see section 3.5).

Reference standard for patients with a positive index test (any combination of):

* tumor cells in cerebrospinal fluid;
* histopathological confirmation (gold standard);
* clinical disease progression during follow-up;
* follow-up MRI diagnostics;
* absence of alpha-fetoprotein (AFP), beta human chorionic gonadotropin (β-hCG) in cerebrospinal fluid or blood.

Reference standard for patients with a negative index test:

• clinical diagnosis of TRb within one year of the last MRI.

The investigators have set a limit of one year for the reference standard of a negative index test to try to avoid patients who develop TRb after the last MRI. The investigators realize that this could falsely classify patients with fast growing tumors that develop after the last MRI, who present with clinical symptoms within a year as true positives. The investigators will evaluate the effect of 'this one year limit' on sensitivity and specificity by varying this limit.

4.1 Secondary objectives After a follow-up period of 5 years survival data will be analyzed. Survival curves will be presented as Kaplan-Meier plots. The log-rank test will be used to compare our date with data from historical patient series. Results will be corrected for potential confounders like differences in treatment, and lead time bias. Stratifications will be made according to tumor size, pineal TRb versus ectropic intracranial TRb, and time between Rb diagnosis and TRb diagnosis.

ELIGIBILITY:
3.2 Inclusion criteria

* All new hereditary and non-hereditary retinoblastoma patients undergoing a baseline MRI diagnosed at one of the ERIC centers.
* Availability of MR sequences (see section 3.7.1) required by the study

We include both hereditary and non-hereditary Rb patients, because it is possible that initially not all patients are classified correctly and because over the course of years, with improving DNA-analysis, more (unilateral) hereditary Rb patients might be detectable (14).

3.3 Exclusion criteria

A patient will be excluded from the study if:

* baseline MRI has not been performed;
* MR protocol or quality not adjusted to the required protocol
* Follow-up not possible or available

When a pineal cyst on baseline MRI is diagnosed, but for some reason no follow-up MRI has been performed, these patients will be specifically followed up to assess its risk of bias and effect on patient survival.

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 3.1 Study population Within ERIC about 150 new retinoblastoma patients are diagnosed every year. About 10 percent of all new retinoblastoma patients will be diagnosed at the VUmc.
Sampling Method: Probability Sample
Enrollment: 607 (Actual)
Dates: Start 2012-10-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of the screening | 01-10-2012
  The sensitivity and specificity of the baseline screening and extended follow-up will be determined

SECONDARY OUTCOMES:
Survival analysis of trilateral retinoblastoma patients | 01-10-2012
  Analysis of (overall) survival after trilateral retinoblastoma

CONTACTS AND LOCATIONS:
Overall Officials: Pim de Graaf, MD PhD, Principal Investigator — Amsterdam UMC
Locations (1):
- VU University Medical Center, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jakobiec FA, Tso MO, Zimmerman LE, Danis P. Retinoblastoma and intracranial malignancy. Cancer. 1977 May;39(5):2048-58. doi: 10.1002/1097-0142(197705)39:53.0.co;2-9. PMID 870165
- [Background] Kivela T. Trilateral retinoblastoma: a meta-analysis of hereditary retinoblastoma associated with primary ectopic intracranial retinoblastoma. J Clin Oncol. 1999 Jun;17(6):1829-37. doi: 10.1200/JCO.1999.17.6.1829. PMID 10561222
- [Background] Rodjan F, de Graaf P, Moll AC, Imhof SM, Verbeke JI, Sanchez E, Castelijns JA. Brain abnormalities on MR imaging in patients with retinoblastoma. AJNR Am J Neuroradiol. 2010 Sep;31(8):1385-9. doi: 10.3174/ajnr.A2102. Epub 2010 Apr 22. PMID 20413604
- [Background] De Potter P, Shields CL, Shields JA. Clinical variations of trilateral retinoblastoma: a report of 13 cases. J Pediatr Ophthalmol Strabismus. 1994 Jan-Feb;31(1):26-31. doi: 10.3928/0191-3913-19940101-06. PMID 8195959
- [Background] Beck Popovic M, Balmer A, Maeder P, Braganca T, Munier FL. Benign pineal cysts in children with bilateral retinoblastoma: a new variant of trilateral retinoblastoma? Pediatr Blood Cancer. 2006 Jun;46(7):755-61. doi: 10.1002/pbc.20464. PMID 16003734
- [Background] Rodjan F, de Graaf P, Brisse HJ, Goricke S, Maeder P, Galluzzi P, Aerts I, Alapetite C, Desjardins L, Wieland R, Popovic MB, Diezi M, Munier FL, Hadjistilianou T, Knol DL, Moll AC, Castelijns JA. Trilateral retinoblastoma: neuroimaging characteristics and value of routine brain screening on admission. J Neurooncol. 2012 Sep;109(3):535-44. doi: 10.1007/s11060-012-0922-4. Epub 2012 Jul 18. PMID 22802019
- [Background] Al-Holou WN, Garton HJ, Muraszko KM, Ibrahim M, Maher CO. Prevalence of pineal cysts in children and young adults. Clinical article. J Neurosurg Pediatr. 2009 Sep;4(3):230-6. doi: 10.3171/2009.4.PEDS0951. PMID 19772406
- [Background] Bossuyt PM, Reitsma JB, Bruns DE, Gatsonis CA, Glasziou PP, Irwig LM, Moher D, Rennie D, de Vet HC, Lijmer JG; Standards for Reporting of Diagnostic Accuracy. The STARD statement for reporting studies of diagnostic accuracy: explanation and elaboration. Clin Chem. 2003 Jan;49(1):7-18. doi: 10.1373/49.1.7. PMID 12507954
- [Background] de Graaf P, Goricke S, Rodjan F, Galluzzi P, Maeder P, Castelijns JA, Brisse HJ; European Retinoblastoma Imaging Collaboration (ERIC). Guidelines for imaging retinoblastoma: imaging principles and MRI standardization. Pediatr Radiol. 2012 Jan;42(1):2-14. doi: 10.1007/s00247-011-2201-5. Epub 2011 Aug 18. PMID 21850471
- [Background] Lacroix-Boudhrioua V, Linglart A, Ancel PY, Falip C, Bougneres PF, Adamsbaum C. Pineal cysts in children. Insights Imaging. 2011 Dec;2(6):671-678. doi: 10.1007/s13244-011-0117-0. Epub 2011 Aug 10. PMID 22347985
- [Background] Pastel DA, Mamourian AC, Duhaime AC. Internal structure in pineal cysts on high-resolution magnetic resonance imaging: not a sign of malignancy. J Neurosurg Pediatr. 2009 Jul;4(1):81-4. doi: 10.3171/2008.5.17681. PMID 19569915